CLINICAL TRIAL: NCT04023786
Title: Positive End-expiratory Pressure Effects to Predict Fluid Responsiveness
Acronym: PEEP-TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-A01599-46
Record Dates: First submitted 2019-07-08; First posted 2019-07-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mechanical Ventilation
Keywords: PEEP test preload dependancy fluid responsiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 70 patients, one arm (Experimental): All patients benefits of a passive leg raising test and a PEEP test to compare these two tests.
  Interventions: Procedure: PEEP-TEST; Device: The VenArt System

INTERVENTIONS:
Procedure: PEEP-TEST — The PEEP test will consist of lowering the PEEP level to 5 cmH2O for a maximum of 2 minutes and a minimum of 1 minute. Patients will be included if the physicians who care for them have decided to set a baseline PEEP level ≥10 cmH2O.
Device: The VenArt System — The VenArt System for estimating cardiac output (a patch stuck to the surface of the neck and a saturation sensor placed at the tip of a finger).

SUMMARY:
Volume expansion is one of the main treatments for shock. A test to predict the effectiveness of volume expansion prior to administration would avoid the need for excess treatment if it proves to be unnecessary.PEEP test would be an easy alternative to the tests used in current practice.

DETAILED DESCRIPTION:
Volume expansion is one of the main treatments for shock, with the goal of increasing cardiac preload and, consequently, cardiac output. However, this increase only occurs if there is a preload-dependence of cardiac output, which is present in 50% of cases. A test to predict the effectiveness of volume expansion prior to administration would avoid the need for excess treatment if it proves to be unnecessary. The end-expiratory pressure test (PEEP) would be to vary the PEEP in patients in shock conditions placed under mechanical ventilation. PEEP is the positive pressure maintained in the airways at the end of expiration. It opposes systemic venous return and lowers cardiac preload. It also distends the pulmonary vessels, increases their resistance and opposes the ejection of the right ventricle. The decrease in PEEP could alleviate the obstacle to venous return and thus increase cardiac preload, mimicking a volume expansion, increasing cardiac output only in the case of preload dependence. This test would be an easy alternative to the tests used in current practice. To evaluate the ability of the PEEP test to detect a preload-dependence condition, defined by a passive passive leg raising test, in patients in shock.

The primary endpoint will be the area under the receiver operating characteristic (ROC) curve constructed to describe the ability of the PEEP test to detect a preload-dependency condition. We measure cardiac output by analysis of the pulse wave contour before and after the passive leg raising and PEEP test tests, then according to these tests, measurement of the cardiac output before and after volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Coverage by a health insurance scheme
  * Patient under mechanical invasive ventilation (tracheal intubation)
  * PEEP level ≥10 cmH2O
  * Cardiac flow monitoring device in place by the PiCCO2 system (Pulsion Medical Systems, Feldkirch, Germany).
  * Ikorus urinary catheter in place
  * Decision by the doctors in charge of carrying out a passive leg raising test and / or a volume expansion

Exclusion Criteria:

* Pregnancy
* Participation in another interventional study
* Patients under the protection of justice
* Thoracic drainage (preventing PEP changes from inducing intrathoracic and transpulmonary pressure changes from their hemodynamic effects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Ability of the PEP test to detect a preload-dependency condition. | At the end of the hospitalization in intensive care unit (1 month maximum)
  The primary endpoint will be the area under the receiver operating characteristic (ROC) curve constructed to describe the ability of the PEP test to detect a preload-dependency condition.

SECONDARY OUTCOMES:
Relationship between the ability of the PEEP test to detect a preload-dependancy and secondly the PEEP delta induced by the test | At the end of the hospitalization in intensive care unit (1 month maximum)
  The secondary endpoint will be the relationship between the area under the curve constructed to describe the ability of the PEP test to detect a preload-dependency state and the PEP delta induced by the test (PEP starting, high, PEP during the test, at 5 cmH2O).
Ability of the PEP test to detect a response to volume expansion. | At the end of the hospitalization in intensive care unit (1 month maximum)
  The secondary endpoint will be the area under the curve constructed to describe the ability of the PEP test to detect a response to volume expansion.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Dr Alexandra Beurton, Le Kremlin-Bicêtre, Val de Marne
  - Dr Alexandra Beurton, Paris

IPD SHARING:
Plan to Share IPD: No